CLINICAL TRIAL: NCT01171742
Title: Effect of Intermittent Hepatic Inflow Occlusion During Donor Hepatectomy In Adult Living Donor Liver Transplantation Using Right Hemiliver Grafts
Brief Title: Effect of Intermittent Hepatic Inflow Occlusion During Donor Hepatectomy In Living Donor Liver Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Samsung Medical Center, JAE WON JOH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-09-096
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: End Stage Liver Disease; Living Donor
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IHIO (Experimental): Intermittent hepatic inflow occlusion (IHIO) by clamping of the portal triad, minimizes blood loss and operation time during liver resection. In addition, ischemic preconditioning with IHIO has been reported to have protective effects in patients undergoing liver resection. IHIO'll be usually performed 3 times during donor liver parenchymal resection, with each IHIO consisting of clamping of the hepatoduodenal ligament for 15 minutes, followed by reperfusion for 5 minutes.
  Interventions: Procedure: Intermittent hepatic inflow occlusion (IHIO)
- Control (Sham Comparator): The donor liver parenchyma'll be transected without IHIO.
  Interventions: Procedure: Intermittent hepatic inflow occlusion (IHIO)

INTERVENTIONS:
Procedure: Intermittent hepatic inflow occlusion (IHIO) — Intermittent hepatic inflow occlusion (IHIO)'ll be usually performed 3 times during donor liver parenchymal resection, with each IHIO consisting of clamping of the hepatoduodenal ligament for 15 minutes, followed by reperfusion for 5 minutes.

SUMMARY:
Intermittent hepatic inflow occlusion (IHIO), also called Pringle maneuver, is a safe and effective procedure for major hepatectomy in patients with liver disease. In addition, ischemic preconditioning with IHIO has been reported to have protective effects in patients undergoing liver resection. The role of IHIO, however, has not been fully elucidated in donors and recipients during living donor liver transplantation.

DETAILED DESCRIPTION:
Intermittent hepatic inflow occlusion (IHIO) by clamping of the portal triad, also called Pringle maneuver, is a safe and effective procedure in major hepatectomy in patients with liver disease. IHIO minimizes blood loss and operation time during liver resection. In addition, ischemic preconditioning with IHIO has been reported to have protective effects in patients undergoing liver resection. In the setting of living donor liver transplantation (LDLT), one of the most important concerns is liver donor safety. Several studies have shown the safety of IHIO in donors for liver transplantation (LT). However, the effect of preconditioning with IHIO during donor hepatectomy on LDLT recipients remains unclear. Several small series have assessed the effects on recipients of ischemic preconditioning during whole liver transplantation from deceased donors. The role of IHIO, however, has not been fully elucidated in liver donors and recipients during LDLT. In this randomized, prospective study, we'll evaluate the efficacy of IHIO in the recipients and donors.

ELIGIBILITY:
Inclusion Criteria:

* Donors and recipient of LDLT, saged ≥18 years, who will undergo LDLT with donors undergoing right hemihepatectomy and recipients receiving right hemiliver grafts
* Informed consent agreement

Exclusion Criteria:

* if the recipients has fulminant hepatic failure
* if the graft to recipient body weight ratio (GRWR) is <0.9
* if a frozen biopsy of the donor liver taken prior to donor hemihepatectomy shows >30% macrovesicular steatosis
* if liver transplantation is ABO incompatible
* if recipients has received previous organ transplants
* if recipients has received or were scheduled to receive multi-organ transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Serum alanine aminotransferase (ALT) concentration within 5 days post-operative | pre-operative and every day till 5 days post-operative
  The primary end-point of this study is peak serum alanine aminotransferase (ALT) concentration within 5 days post-operation on donors and recipients.

SECONDARY OUTCOMES:
post-operative clinical courses, such as liver function tests, hospital stay, and morbidity | During post-operative 1 months or hospitalization
  Secondary end-points in recipients include those involving post-operative clinical courses, such as liver function tests, graft function, stay in the intensive care unit and in-hospital mortality, hospital stay and in donors post-operative clinical courses, such as liver function tests, hospital stay and morbidity requiring additional interveition or delay of hospital stay.
Serum interleukin (IL)-6, IL-8, tumor necrosis factor (TNF)- α, and hepatocyte growth factor (HGF) | In donors immediately after anesthesia induction and 2 hours after graft removal, and in recipients immediately after anesthesia induction, during the anhepatic phase, 2 hours after reperfusion, and at 1 and 3 days post-operatively.
  Blood samples for measurement of interleukin (IL)-6, IL-8, tumor necrosis factor (TNF)- α, and hepatocyte growth factor (HGF) will be taken from donors immediately after anesthesia induction and 2 hours after graft removal, and from recipients immediately after anesthesia induction, during the anhepatic phase, 2 hours after reperfusion, and at 1 and 3 days post-operatively.
Caspase-3 and malondialdehyde in liver biopsy | In donors at the time of laparotomy, just before portal vein and hepatic artery clamping after parenchymal resection, and in recipients two hours after reperfusion
  Biopsy samples'll be taken from donors at the time of laparotomy, just before portal vein and hepatic artery clamping after parenchymal resection, and from recipients two hours after reperfusion. Hepatocyte injury will be determined by measuring the concentrations of caspase-3, and malondialdehyde (MDA) by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Won Joh, MD., PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park JB, Joh JW, Kim SJ, Kwon CH, Chun JM, Kim JM, Moon JI, Lee SK. Effect of intermittent hepatic inflow occlusion with the Pringle maneuver during donor hepatectomy in adult living donor liver transplantation with right hemiliver grafts: a prospective, randomized controlled study. Liver Transpl. 2012 Jan;18(1):129-37. doi: 10.1002/lt.22409. PMID 21837746